CLINICAL TRIAL: NCT01488968
Title: A Phase II Randomized Control Trial of Conventional Versus Hypofractionated Radiation Regimen in Single Phase Using IMRT Technique and Long Term Androgen Suppression Therapy in High-risk Prostate Cancer Patients.
Brief Title: Conventional Versus Hypofractionated Radiation in High Risk Prostate Patients
Acronym: CHIRP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25859
Record Dates: First submitted 2011-12-02; First posted 2011-12-09 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2017-01

CONDITIONS: High-risk Prostate Cancer
Keywords: high risk prostate cancer; hypofractionated radiation treatment; higher biological doses; acceptable rectal toxicity; Radiation Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard (Active Comparator): Standard Radiation Treatment
  Interventions: Radiation: Standard Radiation Treatment
- Hypofractionated (Experimental): Hypofractionated
  Interventions: Radiation: Hypofractionated radiation treatment

INTERVENTIONS:
Radiation: Standard Radiation Treatment — 39 radiation treatments
  Arms: Standard
Radiation: Hypofractionated radiation treatment — 25 radiation treatments
  Arms: Hypofractionated

SUMMARY:
Hypofractionated regimen in high-risk prostate cancer will allow the investigators to deliver higher biological doses to targets in order to improve tumor control and with acceptable rectal toxicity compared to conventional fractionation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient has histologically proven adenocarcinoma of prostate gland by needle core samples or TURP with assigned Gleason score. Prostate biopsy performed within 180 days of enrollment (date of consent).
* Patient has high-risk prostate cancer (stage T3 or T4) and/or PSA greater than or equal to 20 ng/ml and/or Gleason score 8 to 10
* No clinical or radiological evidence of nodal or distant metastasis(es).
* In the opinion of the treating oncologist, patient is fit to undergo radical external beam radiotherapy to the prostate. Patients are accessible for treatment and follow up.
* Patient does not have history of inflammatory bowel disease, anal stenosis, colorectal surgery, or repeated endoscopic examinations/interventions related to anorectal diseases.
* No history of prostatectomy, transurethral resection of prostate on more than one occasion or previous pelvic radiotherapy.
* No history of androgen suppression for greater than or equal to 6 months and patient is willing for androgen suppression treatment as per standard or at physician's discretion.
* No previous malignancy within last five years except BCC or SCC skin or highly curable malignancy where a prognosis for cure is > 80%.
* Patient signed informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-03; Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
The rate of late rectal toxicities between hypofractionated versus conventional fractionated schedules in high risk prostate cancer patients | 5 years

SECONDARY OUTCOMES:
The biochemical control (freedom from PSA failure) rate | 10 years
Disease free survival | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Albert Murtha, Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada